CLINICAL TRIAL: NCT05846061
Title: Epidemiology of Helicobacter Pylori Infection in Children From Slovenia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Tadej Battelino, Professor of paediatrics, University Medical Centre Ljubljana
Other Study IDs: 07011968
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Helicobacter Pylori Infection; Transmission
Keywords: children; infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — stool specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prevalence study population: prevalence study population
  Interventions: Other: Prevalence study population

INTERVENTIONS:
Other: Prevalence study population — No intervention

SUMMARY:
The epidemiology of H. pylori infection among children in Slovenia has not been investigated. Therefore, we are conducting a study to examine the epidemiology of H. pylori and associated risk factors among children in Slovenia.

DETAILED DESCRIPTION:
The population selection was from the three different geographic location in Slovenia. The selection of the studied places was based on their social and economic characteristics and medical provision. We included children from three age groups at the same time we collected information from the parents which may be important for H. pylori transmission.

ELIGIBILITY:
Inclusion Criteria:

* age 6, 14 and 17 years living in three different regions in Slovenia

Exclusion Criteria:

* none

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: children from school of different age groups- community sample
Sampling Method: Non-Probability Sample
Enrollment: 430 (Estimated)
Dates: Start 2021-01-09 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-06-09 (Estimated)

PRIMARY OUTCOMES:
The number of infected children in different age population | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Children's Hospital in Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Polivanova TV, Malaty H, Vshivkov VA. Epidemiology Helicobacter pylori infection in children in the Tyva Republic (Russia). Helicobacter. 2022 Jun;27(3):e12882. doi: 10.1111/hel.12882. Epub 2022 Mar 13. PMID 35285106